CLINICAL TRIAL: NCT01455818
Title: A Multicenter Prospective Cohort Management Study to Evaluate the Safety of Withholding Anticoagulation in Patients With Subsegmental PE Who Have a Negative Serial Bilateral Lower Extremity Ultrasound
Brief Title: A Study to Evaluate the Safety of Withholding Anticoagulation in Patients With Subsegmental PE Who Have a Negative Serial Bilateral Lower Extremity Ultrasound
Acronym: SSPE
Status: Completed | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 2009600-01H
Record Dates: First submitted 2011-10-18; First posted 2011-10-20 (Estimated); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: Subsegmental (Single or Multiple) Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Blood clots in lung arteries (pulmonary embolism) are usually detected using a radiological test called computed tomography (CT scan). As technology advances, the CT scans are able to detect smaller and smaller blood clots. Over time, the frequency of blood clots in the pulmonary arteries has increased significantly (CT scan are now detecting very small blood clots that the investigators could not see before). As a result, more and more people are on blood thinners to treat these small blood clots but their true clinical significance is unknown.

The management of blood thinners is costly and also utilizes scarce healthcare resources. These blood thinners need to be monitored with frequent blood work. Furthermore, every year, approximately 3 percent of patients on blood thinners will have a major bleeding event requiring medical attention.

The investigators don't think that treating these small blood clots in the pulmonary arteries detected on CT scan is worth the risk of bleeding from the blood thinners.

The main goal of this study is to find out if it is safe to not treat very small blood clots in the pulmonary arteries.

The investigators plan to follow 300 patients with small blood clots in their lungs for 90 days. These patients will not be treated with blood thinners but will be followed closely with other non-invasive tests to avoid progression or recurrence of blood clots.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater or equal to 18 years old.
2. Patients with newly diagnosed isolated SSPE* (any number).

   * Isolated SSPE is defined as CTPA demonstrating an intraluminal filling defect in a subsegmental artery with no filling defects visualized at more proximal pulmonary artery levels.

Exclusion Criteria:

1. Proximal lower extremity (popliteal vein or above) or upper extremity (subclavian vein or above) DVT.
2. Need for long term oral anticoagulant therapy for reasons other than VTE.
3. SSPE diagnosed in a hospitalized patient (> 48 hours after hospital admission).
4. Requiring oxygen therapy to maintain an O2 saturation over 92%
5. Previous history of DVT (proximal or distal) of upper or lower extremities, PE, or unusual site thrombosis (e.g. splanchnic or cerebral vein thrombosis).
6. Geographically inaccessible for follow-up
7. Active Malignancy (defined as other than basal-cell or squamous cell carcinoma of the skin; cancer within the past 6 months; any treatment for cancer in the past 6 months; or recurrent or metastatic cancer)
8. Pregnancy
9. Have received more than 48 hours of therapeutic anticoagulation.

   * Prophylactic dose allowed if required for separate indication and acceptable by the investigator.
10. Unable/refuse to sign informed consent
11. Asymptomatic SSPE (e.g. SSPE is an incidental finding on a CT scan conducted for reasons other than suspected PE)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with symptomatic, isolated SSPE* (any number), that are newly diagnosed by computed tomographic pulmonary angiography will be eligible to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 292 (Actual)
Dates: Start 2011-03; Primary Completion 2021-03 (Actual); Study Completion 2021-05 (Actual)

PRIMARY OUTCOMES:
Recurrent VTE | 90 day follow-up
  Recurrent VTE will be diagnosed according to previously published criteria: 1)Lower extremity US revealing non-compressibility at the trifurcation of the popliteal vein or above; OR 2) Venography demonstrating a constant intraluminal filling defect above the trifurcation of the popliteal vein; OR 3) Pulmonary angiography demonstrating a new constant intraluminal filling defect or a cut off of a vessel; OR 4) Ventilation/perfusion scanning with a high probability of PE; OR 5) CTPA demonstrating new intraluminal filling defect in a subsegmental or greater sized pulmonary artery; OR 6) PE discovered at autopsy.

SECONDARY OUTCOMES:
Interobserver agreement for SSPE diagnosis on CTPA (local Vs. central interpretation) | 90 day follow-up
Death due to PE | 90 day follow-up
  Definition of death due to PE Certain: hypotension, hypoxia, cardiac arrest with no other explanation other than PE and autopsy or radiographic confirmation Highly probable: criteria for certain but another disease could have caused the death Probable: other cause suspected based on clinical evidence but 100% certainty not available Unlikely: all other cases
Death probably due to PE | 90 day follow-up
  Certain: hypotension, hypoxia, cardiac arrest with no other explanation other than PE and autopsy or radiographic confirmation Highly probable: criteria for certain but another disease could have caused the death Probable: other cause suspected based on clinical evidence but 100% certainty not available Unlikely: all other cases
Major bleeding | 90 day follow-up
  Major bleeding will be defined according to previously published criteria (51):
  1. Fatal bleeding; OR
  2. Symptomatic bleeding in a critical area or organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intraarticular or pericardial, or intramuscular with compartment syndrome; OR
  3. Bleeding causing a fall in hemoglobin level of 20 g/L (1.24 mmol/L) or more, or leading to transfusion of two or more units of whole blood or red cells
Minor bleeding | 90 day follow-up
  Minor bleeding will be defined as any bleeding not meeting the requirements of a major bleeding event.

CONTACTS AND LOCATIONS:
Locations (9):
- Canada (7):
  - Capital District Health Authority, Halifax, Nova Scotia
  - Hamilton General Hospital, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - Ottawa Hospital, Ottawa, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Sir Mortimer B. Davis Jewish General Hospital, Montreal, Quebec
  - St. Mary's Hospital Centre, Montreal, Quebec
- Centre Hospitalier Universitaire de Brest, Brest, France
- Geneva Hospital, Geneva, Switzerland

REFERENCES:
- [Derived] Le Gal G, Kovacs MJ, Bertoletti L, Couturaud F, Dennie C, Hirsch AM, Huisman MV, Klok FA, Kraaijpoel N, Mallick R, Pecarskie A, Pena E, Phillips P, Pichon I, Ramsay T, Righini M, Rodger MA, Roy PM, Sanchez O, Schmidt J, Schulman S, Shivakumar S, Trinh-Duc A, Verdet R, Vinsonneau U, Wells P, Wu C, Yeo E, Carrier M; SSPE Investigators. Risk for Recurrent Venous Thromboembolism in Patients With Subsegmental Pulmonary Embolism Managed Without Anticoagulation : A Multicenter Prospective Cohort Study. Ann Intern Med. 2022 Jan;175(1):29-35. doi: 10.7326/M21-2981. Epub 2021 Nov 23. PMID 34807722